CLINICAL TRIAL: NCT06263621
Title: Changing Restaurant Portion Size Descriptions to Encourage Selection and Intake of Smaller Meals: a Field Experiment
Brief Title: Changing Portion Size Descriptions in a Cafeteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Restaurant Associates (Unknown)
Responsible Party: Principal Investigator, Sophia Hua, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 855090
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Food Selection; Obesity; Weight Gain; Food Preferences
Keywords: portion size, choice behavior, energy intake, food labeling
MeSH Terms: conditions — Food Preferences; Obesity; Weight Gain

STUDY DESIGN:
Intervention Model Description: Entrees are offered in two different portion sizes at two cafes. The cafes were randomized to either receive the "Standard" portion label for the smaller size (Intervention) or the "Small" portion label for the smaller size (Control). The larger portion was labeled "Large." Daily lunch transaction data will be provided by the cafes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention "Standard" (Experimental): The smaller entree is labeled "Standard" and the larger entree is labeled "Large."
  Interventions: Behavioral: Intervention "Standard"
- Control "Small" (No Intervention): The smaller entree is labeled "Small" and the larger entree is labeled "Large."

INTERVENTIONS:
Behavioral: Intervention "Standard" — The two cafes will offer entrees in two sizes, a smaller and larger size. In the intervention cafe, the smaller size will be labeled "Standard" during the intervention period, and "Small" during all other times. In the control cafe, the smaller size will always be labeled "Small." The larger size will always be labeled "Large" for both cafes during the duration of the study.
  Other Names: "Standard"
  Arms: Intervention "Standard"

SUMMARY:
The goal of this this intervention is to test the degree to which a portion size labeling intervention influences consumer selection of smaller portions at two large cafés. The main question it aims to answer is: Do consumers order fewer calories when the portion size label for the smaller entree is called "standard" instead of "small"?

Participants will order lunch as usual in the two cafes (one intervention, one control) for 5.5 months, and all order items will be recorded in the check-out system. One cafe will receive the labeling intervention, while the other will not. Researchers will compare the average calories per order between the two cafes to see if there are differences.

DETAILED DESCRIPTION:
The investigators will work with two cafés that will start offering two size options for their entrées. The cafés will go through three phases: a baseline phase where there are two portion sizes and no intervention (6 weeks), an intervention phase where the portion size labeling strategy will be implemented (7 weeks), and then a final phase where the portion size intervention is removed (7 weeks). During the baseline period, the smaller-sized entrée will not receive a label, and the larger-sized entrée will be called "Large." During the intervention period for the control café, labeling will stay the same, but in the intervention café, the smaller size will be labeled "Standard" and the larger size will be called "Large." In the post-intervention period, the smaller-sized entrée in the intervention café will have no label so that it resembles the control café.

ELIGIBILITY:
Inclusion Criteria:

* All customers who make a lunch purchase at the cafes

Exclusion Criteria:

* Purchases made outside of lunch service.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 101481 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Average kcal per entree sold | Daily sales data for 5.5 months
  The primary outcome will be the average kcal per entrée purchased.

SECONDARY OUTCOMES:
Number of entrée units purchased | Daily sales data for 5.5 months
  Analyzing the number of entrée units purchased will enable the investigators to assess the impact of the intervention on entree sales.
Total kcal per transaction | Daily sales data for 5.5 months
  This will allow the investigators to examine whether participants who ordered a reduced-sized entrée were ordering more calories in other parts of the meal (i.e., a dessert).
Weekly gross sales | Daily sales data for 5.5 months
  This will allow the investigators to assess whether the addition of a reduced-sized entrée at a lower cost negatively affected lunch service revenue.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia V Hua, PhD, MPH, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Courtyard Cafe, Boston, Massachusetts
  - Elements Cafe, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided
Sales data will be made available to interested researchers pending approval from cafe managers.